CLINICAL TRIAL: NCT02444065
Title: Rapid Response to Day Hospital Treatment in Bulimia Nervosa and Purging Disorder: A Randomized Controlled Trial of an Intervention to Facilitate Early Symptom Change
Brief Title: Rapid Response to Day Hospital Treatment in Bulimia Nervosa and Purging Disorder
Acronym: CBT-RR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-7391-B
Record Dates: First submitted 2015-04-23; First posted 2015-05-14 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Bulimia Nervosa; Eating Disorder
Keywords: Cognitive behavior therapy; Motivational interviewing; Bulimia nervosa; Rapid response
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders | interventions — Cognitive Behavioral Therapy; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavior Therapy (CBT) (Experimental): In this arm, participants receive the Cognitive behavior therapy (CBT) intervention as an augmentative treatment to standard day hospital treatment as usual.
  Interventions: Behavioral: Cognitive Behavior Therapy (CBT)
- Motivational Interviewing (MI) (Active Comparator): In this arm, participants receive the Motivational Interviewing intervention as an augmentative treatment to standard day hospital treatment as usual.
  Interventions: Behavioral: Motivational Interviewing (MI)

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy (CBT) — The CBT intervention is a 4 session (1 hour each) individual psychotherapy intervention that uses a manualized treatment protocol developed by the investigators. It uses standard CBT for eating disorders interventions, including orientation to the CBT model, psychoeducation, commitment and goal setting, behavioral strategies for normalizing eating and reducing bulimic symptoms, planning, and homework. 1-2 sessions are delivered before starting day hospital treatment, and the remaining sessions are delivered in the first weeks of day hospital.
  Arms: Cognitive Behavior Therapy (CBT)
Behavioral: Motivational Interviewing (MI) — The MI intervention is a 4 session (1 hour each) individual psychotherapy intervention that uses a manualized treatment protocol (Carter & Bewell-Weiss, 2012). It uses standard MI for eating disorders interventions, including decisional balance, exploring values, readiness and confidence rules, and MI communication strategies. 1-2 sessions are delivered before starting day hospital treatment, and the remaining sessions are delivered in the first weeks of day hospital.
  Arms: Motivational Interviewing (MI)

SUMMARY:
Treatments for bulimia nervosa (BN) have relatively high rates of nonremission and relapse, meaning that improving treatments is a high priority in this area. Rapid response to treatment -cessation of binge eating and vomiting symptoms within the first weeks of treatment - is a robust predictor of improved post-treatment outcomes and lower relapse rates, but no study has tried to facilitate rapid response as a means of improving treatment outcomes. The present study responds to this gap in the literature by testing a 4-session CBT-based individual intervention for rapid response (i.e., "CBT-RR"), designed to augment standard day hospital (DH) treatment for BN and Purging Disorder (PD) by focusing on strategies and skills for rapid symptom interruption. CBT-RR will be compared to a matched-intensity augmentative motivational interviewing (MI) intervention. Participants will be recruited from a hospital-based day program for eating disorders, and will be randomly assigned to one of the two conditions in addition to the DH as usual. participants will be assessed at pre-intervention, post-intervention, week 4 of DH, post-DH, and 6 months follow-up. It is hypothesized that compared to those who receive MI, patients who receive CBT-RR will be more likely to exhibit a rapid response to day hospital treatment (i.e., </= 3 binge eating and/or vomiting episodes in the first 4 weeks). It is further hypothesized that patients who receive CBT-RR will exhibit fewer binge eating and/or vomiting episodes at post-DH and at 6-month follow-up. Potential mediators and moderators of these hypothesized treatment effects will be examined on an exploratory basis, including self-efficacy, motivation, and hope (potential mediators), and emotion regulation, depression, cognitive psychopathology of eating disorders, and working alliance with the therapist (potential moderators).

DETAILED DESCRIPTION:
Cognitive behaviour therapy (CBT) is the most empirically supported treatment for bulimia nervosa (BN) and related disorders, yet approximately 1/3 of completers do not remit, there is a substantial treatment attrition rate, and 1/3 of remitted patients will relapse within the first 2 years. Improving CBT is an important research prerogative. Motivational interviewing (MI) is an augmentative intervention that has been investigated to improve CBT, but reviews indicate that it is not efficacious with eating disorders. The failure of MI with eating disorders has led to consideration that focusing on early behaviour change might be a more productive therapeutic strategy. Rapid response to treatment for eating disorders has been reliably identified as a prognostic indicator in eating disorders. For BN and similar disorders, rapid response is the rapid reduction of binge eating, vomiting, and dietary restriction during the first few weeks of treatment. Numerous studies have indicated that patients who rapidly respond to treatment are significantly more likely to be remitted at post treatment and significantly less likely to relapse, compared to those who respond more slowly. No preexisting clinical, demographic, personality or other factors have clearly emerged to account for this effect. Given that rapid response has clear prognostic importance, and given that research has failed to identify mechanisms driving this finding, this study seeks to determine whether rapid response can be facilitated clinically using a targeted intervention designed to provide patients with specific behavioural skills to decrease their bulimic symptoms rapidly. Improving remission and relapse rates is a high priority in the eating disorders research field. the investigators already know that cognitive and behavioural strategies have efficacy for eating disorders, but existing treatments need improvement. Rapid response is an area that has been frequently described and has clear prognostic importance and no clear mechanism accounting for why some patients rapidly respond, suggesting that perhaps rapid response could be facilitated if patients are provided with the skills, mindset, and support to do so. However, no study to date has sought to answer this question and determine whether rapid response can be facilitated in order to improve patient prognoses. Thus, this study seeks to examine whether rapid response to day hospital treatment can be facilitated clinically using an augmentative CBT based intervention targeting early symptom change. The CBT intervention will be compared to a matched-intensity motivational interviewing (MI) intervention. The rationale for using MI is because MI is frequently used to augment standard treatments, it provides an active treatment comparison, and because the rationale for the present study emerged partly from research aimed at understanding some of the limitations of MI in treating eating disorders. Thus, MI provides a theoretically-driven comparison group. It is predicted that individuals who receive CBT (versus MI) will be more likely to be classified as rapid responders, and will have fewer bulimic symptoms at post-day hospital and 6-month follow-up. As well, it is hypothesized that changes in self-efficacy, motivation, or hopefulness may help to account for these findings.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bulimia nervosa or other specified feeding and eating disorder (OSFED) purging disorder
* Body mass index of 19.0 or higher
* Has accepted day hospital eating disorder treatment at the Toronto General Hospital Eating Disorder Day Hospital Program
* No previous treatments at the Toronto General Hospital Eating Disorder Day Hospital Program in the previous 5 years
* Can read and write English fluently.

Exclusion Criteria:

* Current imminent suicidality
* Current manic episode
* Current psychosis
* Current medical instability as assessed by program medical team.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Rapid response to day hospital treatment | First 4 weeks of day hospital treatment
  Rapid response is a binary outcome variable (yes/no) of early bulimic symptoms. Rapid responders exhibit a total of three or fewer binge and/or vomit and/or laxative episodes in the first four weeks of day hospital treatment for eating disorders.
Changes in bulimic symptom frequency | Each of the following: Baseline, first 4 weeks of day hospital, last 4 weeks of day hospital, and months 1-6 in follow-up.
  Bulimic symptoms (binge eating and/or vomiting and/or laxative use) will be totalled for each 4 week period and changes modelled over time at the following time points: Baseline, first 4 weeks of day hospital, last 4 weeks of day hospital, and months 1-6 in follow-up.

SECONDARY OUTCOMES:
End-of-Day Hospital Outcome | Participants will be assessed at end of day hospital stay, an expected average of 8 weeks.
  Outcome is a binary outcome variable, remitted (yes/no). Remitted patients have one or fewer binge and/or vomit and/or laxative episodes in the last 4 weeks of day hospital treatment. Non-remitted patients have 2 or more episodes in this same period. Day hospital stays are expected to consist of an average of 8 weeks of treatment.
6-month relapse rate | 6 months after discharge from day hospital
  Relapse is a binary outcome variable (yes/no). Relapsed patients have an average of 4 or more binge and/or vomit and/or laxative use episodes per month for three consecutive months, beginning in the first 6 months after discharge from day hospital program. Non-relapsed patients have bulimic symptoms below this threshold.

OTHER OUTCOMES:
Self-Efficacy | Each of the following: Baseline, Session 2 (on average the week before starting Day Hospital or Day Hospital week 1), Day Hospital Week 4, End of Day hospital (average=8 weeks)
  Changes in self-efficacy will be modelled across several time points (baseline, session 2, week 4 of day hospital, and post-day hospital). Changes in self-efficacy from baseline to the 4th week in day hospital treatment will also be examined as a potential mediator of the effects of treatment on rapid response. Self-efficacy will be measured using the Readiness and Motivation Questionnaire (Geller et al., 2013). Day hospital stays are expected to consist of an average of 8 weeks of treatment.
Motivation | Each of the following: Baseline, Session 2 (on average the week before starting Day Hospital or Day Hospital week 1), Day Hospital Week 4, End of Day hospital (average=8 weeks)
  Changes in motivation will be modelled across several time points (baseline, session 2, week 4 of day hospital, and post-day hospital). Changes in motivation from baseline to the 4th week in day hospital treatment will also be examined as a potential mediator of the effects of treatment on rapid response. Motivation will be measured using the Readiness and Motivation Questionnaire (Geller et al., 2013). Day hospital stays are expected to consist of an average of 8 weeks of treatment.
Hope | Each of the following: Baseline, Session 2 (on average the week before starting Day Hospital or Day Hospital week 1), Day Hospital Week 4, End of Day hospital (average=8 weeks)
  Changes in hope will be modelled across several time points (baseline, session 2, week 4 of day hospital, and post-day hospital). Changes in hope from baseline to the 4th week in day hospital treatment will also be examined as a potential mediator of the effects of treatment on rapid response. Hope will be measured using an investigator-constructed questionnaire. Day hospital stays are expected to consist of an average of 8 weeks of treatment.
Moderator of treatment response - emotion regulation | Baseline
  Emotion regulation skills at baseline will be examined as a potential moderator of treatment response.
Moderator of treatment response - depression symptoms | Baseline
  Depression symptoms at baseline will be examined as a potential moderator of treatment response.
Moderator of treatment response - weight-based self-esteem | Baseline
  Weight-based self-esteem at baseline will be examined as a potential moderator of treatment response.
Moderator of treatment response - working alliance with the therapist | Week 4
  Working alliance with study therapist will be examined as a potential moderator of treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Traci McFarlane, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Eating Disorder Program, Toronto, Ontario, Canada

REFERENCES:
- [Background] Macdonald P, Hibbs R, Corfield F, Treasure J. The use of motivational interviewing in eating disorders: a systematic review. Psychiatry Res. 2012 Nov 30;200(1):1-11. doi: 10.1016/j.psychres.2012.05.013. Epub 2012 Jun 18. PMID 22717144
- [Result] Agras WS, Crow SJ, Halmi KA, Mitchell JE, Wilson GT, Kraemer HC. Outcome predictors for the cognitive behavior treatment of bulimia nervosa: data from a multisite study. Am J Psychiatry. 2000 Aug;157(8):1302-8. doi: 10.1176/appi.ajp.157.8.1302. PMID 10910795
- [Result] Bulik CM, Sullivan PF, Carter FA, McIntosh VV, Joyce PR. Predictors of rapid and sustained response to cognitive-behavioral therapy for bulimia nervosa. Int J Eat Disord. 1999 Sep;26(2):137-44. doi: 10.1002/(sici)1098-108x(199909)26:23.0.co;2-n. PMID 10422602
- [Result] Wilson GT, Fairburn CC, Agras WS, Walsh BT, Kraemer H. Cognitive-behavioral therapy for bulimia nervosa: time course and mechanisms of change. J Consult Clin Psychol. 2002 Apr;70(2):267-74. PMID 11952185
- [Result] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Bohn K, Hawker DM, Wales JA, Palmer RL. Transdiagnostic cognitive-behavioral therapy for patients with eating disorders: a two-site trial with 60-week follow-up. Am J Psychiatry. 2009 Mar;166(3):311-9. doi: 10.1176/appi.ajp.2008.08040608. Epub 2008 Dec 15. PMID 19074978
- [Result] Grilo CM, Masheb RM. Rapid response predicts binge eating and weight loss in binge eating disorder: findings from a controlled trial of orlistat with guided self-help cognitive behavioral therapy. Behav Res Ther. 2007 Nov;45(11):2537-50. doi: 10.1016/j.brat.2007.05.010. Epub 2007 Jun 7. PMID 17659254
- [Result] McFarlane TL, MacDonald DE, Royal S, Olmsted MP. Rapid and slow responders to eating disorder treatment: a comparison on clinically relevant variables. Int J Eat Disord. 2013 Sep;46(6):563-6. doi: 10.1002/eat.22136. Epub 2013 Apr 12. PMID 23580395
- [Result] Knowles L, Anokhina A, Serpell L. Motivational interventions in the eating disorders: what is the evidence? Int J Eat Disord. 2013 Mar;46(2):97-107. doi: 10.1002/eat.22053. Epub 2012 Sep 24. PMID 23001832
- [Result] MacDonald DE, Trottier K, McFarlane T, Olmsted MP. Empirically defining rapid response to intensive treatment to maximize prognostic utility for bulimia nervosa and purging disorder. Behav Res Ther. 2015 May;68:48-53. doi: 10.1016/j.brat.2015.03.007. Epub 2015 Mar 17. PMID 25800137
- [Result] Masheb RM, Grilo CM. Rapid response predicts treatment outcomes in binge eating disorder: implications for stepped care. J Consult Clin Psychol. 2007 Aug;75(4):639-44. doi: 10.1037/0022-006X.75.4.639. PMID 17663617
- [Result] McFarlane T, Olmsted MP, Trottier K. Timing and prediction of relapse in a transdiagnostic eating disorder sample. Int J Eat Disord. 2008 Nov;41(7):587-93. doi: 10.1002/eat.20550. PMID 18473336
- [Result] Olmsted MP, Kaplan AS, Rockert W. Rate and prediction of relapse in bulimia nervosa. Am J Psychiatry. 1994 May;151(5):738-43. doi: 10.1176/ajp.151.5.738. PMID 8166317
- [Result] Olmsted MP, Kaplan AS, Rockert W, Jacobsen M. Rapid responders to intensive treatment of bulimia nervosa. Int J Eat Disord. 1996 Apr;19(3):279-85. doi: 10.1002/(SICI)1098-108X(199604)19:33.0.CO;2-J. PMID 8704727
- [Result] Olmsted MP, MacDonald DE, McFarlane T, Trottier K, Colton P. Predictors of rapid relapse in bulimia nervosa. Int J Eat Disord. 2015 Apr;48(3):337-40. doi: 10.1002/eat.22380. Epub 2014 Dec 26. PMID 25545720
- [Result] Olmsted MP, McFarlane T, Trottier K, Rockert W. Efficacy and intensity of day hospital treatment for eating disorders. Psychother Res. 2013;23(3):277-86. doi: 10.1080/10503307.2012.721937. Epub 2012 Sep 18. PMID 22989039
- [Result] Raykos BC, Watson HJ, Fursland A, Byrne SM, Nathan P. Prognostic value of rapid response to enhanced cognitive behavioral therapy in a routine clinic sample of eating disorder outpatients. Int J Eat Disord. 2013 Dec;46(8):764-70. doi: 10.1002/eat.22169. Epub 2013 Aug 5. PMID 23913536
- [Result] Thompson-Brenner H, Shingleton RM, Sauer-Zavala S, Richards LK, Pratt EM. Multiple measures of rapid response as predictors of remission in cognitive behavior therapy for bulimia nervosa. Behav Res Ther. 2015 Jan;64:9-14. doi: 10.1016/j.brat.2014.11.004. Epub 2014 Nov 13. PMID 25462877
- [Result] Vaz AR, Conceicao E, Machado PP. Early response as a predictor of success in guided self-help treatment for bulimic disorders. Eur Eat Disord Rev. 2014 Jan;22(1):59-65. doi: 10.1002/erv.2262. Epub 2013 Oct 4. PMID 24123526
- [Result] Waller G. The myths of motivation: time for a fresh look at some received wisdom in the eating disorders? Int J Eat Disord. 2012 Jan;45(1):1-16. doi: 10.1002/eat.20900. Epub 2011 Feb 14. PMID 22170018
- [Result] Zunker C, Peterson CB, Cao L, Mitchell JE, Wonderlich SA, Crow S, Crosby RD. A receiver operator characteristics analysis of treatment outcome in binge eating disorder to identify patterns of rapid response. Behav Res Ther. 2010 Dec;48(12):1227-31. doi: 10.1016/j.brat.2010.08.007. Epub 2010 Sep 6. PMID 20869041
- [Result] Zeeck A, Weber S, Sandholz A, Wetzler-Burmeister E, Wirsching M, Hartmann A. Inpatient versus day clinic treatment for bulimia nervosa: a randomized trial. Psychother Psychosom. 2009;78(3):152-60. doi: 10.1159/000206869. Epub 2009 Mar 9. PMID 19270470
- [Result] Begin C, Gagnon-Girouard MP, Aime A, Ratte C. Trajectories of eating and clinical symptoms over the course of a day hospital program for eating disorders. Eat Disord. 2013;21(3):249-64. doi: 10.1080/10640266.2013.779188. PMID 23600555
- [Result] Byrne SM, Fursland A, Allen KL, Watson H. The effectiveness of enhanced cognitive behavioural therapy for eating disorders: an open trial. Behav Res Ther. 2011 Apr;49(4):219-26. doi: 10.1016/j.brat.2011.01.006. Epub 2011 Jan 27. PMID 21345418
- [Result] Horvath, A. O., & Greenberg, L. S. (1989). Development and validation of the Working Alliance Inventory. Journal of Counselling Psychology, 36, 223-233. doi:10.1037/0022-0167.36.2.223
- [Result] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). Beck Depression Inventory-II. San Antonio, TX: Pearson.
- [Result] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54. doi:10.1007/s10862-008-9102-4
- [Result] Geller J, Brown KE, Srikameswaran S, Piper W, Dunn EC. The psychometric properties of the Readiness and Motivation Questionnaire: a symptom-specific measure of readiness for change in the eating disorders. Psychol Assess. 2013 Sep;25(3):759-768. doi: 10.1037/a0032539. Epub 2013 May 6. PMID 23647034
- [Result] Trottier K, McFarlane T, Olmsted MP, McCabe RE. The Weight Influenced Self-Esteem Questionnaire (WISE-Q): factor structure and psychometric properties. Body Image. 2013 Jan;10(1):112-20. doi: 10.1016/j.bodyim.2012.08.008. Epub 2012 Oct 12. PMID 23068567